CLINICAL TRIAL: NCT01342341
Title: Placebo-Controlled Cross Over Trial of Chlorzoxazone Intake
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Chlorzoxazone
Record Dates: First submitted 2011-04-19; First posted 2011-04-27 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism | interventions — Chlorzoxazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parafon Forte first, then Placebo (Experimental): Experimental: Forty moderate to heavy social alcohol users (women=10-25 drinks/week, men=14-30 drinks/week) will receive either 250 or 500 mg of chlorzoxazone BID (500 or 1000 mg/day) x 7 days followed by 500 or 1000 mg of chlorzoxazone BID (1000 or 2000 mg/day) x 7 days (1st intervention; 14 days), followed by a washout (7 days), and then followed by placebo (2nd intervention; 14 days).
  Interventions: Drug: Parafon Forte
- Placebo first, then Parafon Forte (Placebo Comparator): Experimental: Forty moderate to heavy social alcohol users (women=10-25 drinks/week, men=14-30 drinks/week) will receive placebo (1st intervention; 14days) followed by a washout (7 days), and then followed by either 250 or 500 mg of chlorzoxazone BID (500 or 1000 mg/day) x 7 days followed by 500 or 1000 mg of chlorzoxazone BID (1000 or 2000 mg/day) x 7 days (2nd intervention; 14 days).
  Interventions: Drug: Parafon Forte

INTERVENTIONS:
Drug: Parafon Forte — Drug: Parafon Forte administered at study visit
  Other: Placebo administered at study visit
  Other Names: Chlorzoxazone

SUMMARY:
The overall goals of this study are to (1) expand knowledge about interactions of chlorzoxazone with alcohol by assessing the effects of chlorzoxazone compared to placebo in moderate and heavy social alcohol users and (2) to compare the effects of chlorzoxazone on visual cue induced alcohol craving to placebo in moderate to heavy social alcohol users.

DETAILED DESCRIPTION:
The investigators propose a 45-day, double-blind, placebo-controlled crossover study in light to moderate and heavy alcohol users.

The specific aims are to:

1. Determine if chlorzoxazone alters daily alcohol consumption by comparing the mean drinks consumed per day during chlorzoxazone administration compared with the mean drinks per day consumed during placebo administration.
2. To determine if polymorphisms in genes encoding for neurotransmitters or receptors involved in alcohol reward, abuse, dependence, craving, or relapse may predict the level of response to chlorzoxazone's effects on alcohol consumption or craving.
3. To investigate any change in alcohol craving during a cue induced craving task where participants view and respond to a number of images.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria: Healthy adults who are social drinkers 21 - 50 years of age.

1. Moderate to heavy social drinkers (women=10-25 drinks/week, men=14-30 drinks/week).
2. If female, must be non-lactating, not pregnant, and using a reliable contraception method (i.e. abstinence, intrauterine device [IUD], or hormonal birth control).
3. Able and willing to provide written informed consent.
4. Able to understand and follow the instructions of the investigator, and understand all rating scales.

Exclusion Criteria:

1. Use of cocaine, amphetamines, hallucinogens, "ecstasy", opiates, sedatives, pain pills, sleeping pills, or other psychoactive drugs more than twice a week.
2. A history of complicated alcohol or other drug withdrawal syndrome(s), e.g. delirium tremens or seizures.
3. Current physiological dependence on any psychoactive drug (except nicotine or caffeine) including alcohol, as determined by MD or NP assessment.
4. Current enrollment in an alcohol or other drug treatment program, or current legal problems relating to alcohol or other drug use, including awaiting trial or supervision by a parole or probation officer.
5. Currently trying to quit using alcohol and/or "recreational" drugs.
6. Clinically significant medical or psychiatric illness as determined by screening blood tests, medical history, and physical exam performed or reviewed by the study MD or NP.
7. Bilirubin more than 2 times the normal upper limit.
8. AST (SGOT), ALT (SGPT), or alkaline phosphatase more than 2 ½ times the normal upper limit.
9. Symptoms of liver disease, as assessed by MD or NP assessment (jaundice, Hx of hepatitis, itchy skin, etc.).
10. A current pregnancy, or a woman of child-bearing potential not currently using an adequate means of contraception.
11. BAC level greater than 0.05% at the beginning of Screening Visit, Visit 1 or Visit 4.
12. Neurological dysfunction or psychiatric disorder severe enough to interfere with assessment of outcome measures as defined above.
13. Known allergy to chlorzoxazone.
14. Has received an investigational drug within 30 days prior to Study Visit 2 (after screening visit).
15. Subjects who are unable to read or speak English.
16. Those who, in the opinion of the investigator, are considered unable to adhere to scheduled appointments, are unlikely to comply with the study protocol, or who are unsuitable for any other reason.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Fields, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Ernest Gallo Clinic and Research Center, Emeryville, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Parafon Forte First, Then Placebo: Participants will receive either 250 or 500 mg of chlorzoxazone BID (500 or 1000 mg/day) x 7 days followed by 500 or 1000 mg of chlorzoxazone BID (1000 or 2000 mg/day) x 7 days (1st intervention; 14 days), followed by a washout (7 days), and then followed by placebo (2nd intervention; 14 days).
- Placebo First, Then Parafon Forte: Participants will receive placebo (1st intervention; 14days) followed by a washout (7 days), and then followed by either 250 or 500 mg of chlorzoxazone BID (500 or 1000 mg/day) x 7 days followed by 500 or 1000 mg of chlorzoxazone BID (1000 or 2000 mg/day) x 7 days (2nd intervention; 14 days).
Period: Overall Study
Arm/Group | Parafon Forte First, Then Placebo | Placebo First, Then Parafon Forte
Started | 24 | 24
Completed | 20 | 20
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parafon Forte First, Then Placebo | Placebo First, Then Parafon Forte | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Consumption in Drinks/Week.
Description: Each subject will record how many drinks/week they are consuming while on the study drug and placebo during the 45-day study. The primary outcome of this study is to determine the effect of chlorzoxazone on alcohol consumption. Reduction in alcohol consumption is measured utilizing behavioral inventories, electronic diaries, urine, and ethyl glucuronide.
Time Frame: 45 days
Measure: Mean (Standard Deviation); unit: number of drinks
Groups:
- Parafon Forte: Participants received either 250 or 500 mg of chlorzoxazone BID (500 or 1000 mg/day) x 7 days followed by 500 or 1000 mg of chlorzoxazone BID (1000 or 2000 mg/day) x 7 days (1st intervention; 14 days), followed by a washout (7 days), and then followed by placebo (2nd intervention; 14 days).
- Placebo: Participants received placebo (1st intervention; 14 days) followed by a washout (7 days), and then followed by either 250 or 500 mg of chlorzoxazone BID (500 or 1000 mg/day) x 7 days followed by 500 or 1000 mg of chlorzoxazone BID (1000 or 2000 mg/day) x 7 days (2nd intervention; 14 days).
Arm/Group | Parafon Forte | Placebo
Number analyzed (Participants) | 40 | 40
number of drinks | 83.43 (55.65) | 75.97 (42.16)

ADVERSE EVENTS:
Time Frame: From enrollment through study completion, up to 45 days
Groups:
- Parafon Forte: This is a cross-over study. Adverse Events Arms/Groups are reported "per intervention". Group reflects **all** participants who received Parafon Forte intervention during the study.
- Placebo: This is a cross-over study. Adverse Events Arms/Groups are reported "per intervention". Group reflects **all** participants who received Placebo intervention during the study.
Arm/Group | Parafon Forte | Placebo
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No